CLINICAL TRIAL: NCT03005145
Title: Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness: Randomized Controlled Trial
Brief Title: Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0796
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2023-11

CONDITIONS: Bacteremia; Intensive Care; Critically Ill; Sepsis; Mortality; Antimicrobial
MeSH Terms: conditions — Bacteremia; Critical Illness; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short duration (7 days) (Active Comparator): Patients in 7 day arm will receive adequate antibiotics until the end of day 7 only
  Interventions: Other: 7 days of adequate antibiotic treatment
- Long duration (14 days) (Active Comparator): Patients in 14 day arm will receive adequate antibiotics until the end of day 14 only
  Interventions: Other: 14 days of adequate antibiotic treatment.

INTERVENTIONS:
Other: 7 days of adequate antibiotic treatment — The choice of treatment including type, dose, route and interval of antibiotic will be left at the discretion of treating team as long as it is appropriate for the bacteremia
  Arms: Short duration (7 days)
Other: 14 days of adequate antibiotic treatment. — The choice of treatment including type, dose, route and interval of antibiotic will be left at the discretion of treating team as long as it is appropriate for the bacteremia
  Arms: Long duration (14 days)

SUMMARY:
The World Health Organization, U.S. Centers for Disease Control and Prevention, Association of Medical Microbiology and Infectious Diseases (AMMI) Canada, and Health Canada have all declared antimicrobial resistance a global threat to health, based on rapidly increasing resistance rates and declining new drug development. Up to 30-50% of antibiotic use is inappropriate, and excessive durations of treatment are the greatest contributor to inappropriate use. Shorter duration treatment (≤7 days) has been shown in meta-analyses to be as effective as longer antibiotic treatment for a range of mild to moderate infections. A landmark trial in critically ill patients with ventilator-associated pneumonia showed that mortality and relapse rates were non-inferior in patients who received 8 vs 15 days of treatment. Similar adequately powered randomized trial evidence is lacking for the treatment of patients with bloodstream infections caused by a wide spectrum of organisms.

DETAILED DESCRIPTION:
Bloodstream infections are a common and serious problem, increasing length of hospital stay by 2-3 weeks, adding $25,000-40,000 in excess hospital costs, and tripling the risk of death. At the same time, antibiotic overuse is also a common and serious problem, in that 30-50% of antibiotic use is unnecessary or inappropriate, and results in avoidable drug side effects such as kidney failure, Clostridioides difficile infection, increased costs, and spiralling antibiotic resistance rates. The greatest contributor to antibiotic overuse is excessive durations of treatment.

Extensive research has demonstrated that shorter duration antibiotic treatment (less or equal to 7 days) is as effective as longer duration treatment for a variety of infectious diseases, but this question has not been directly studied in the setting of bloodstream infection. BALANCE team's systematic review of the medical literature, national survey of Canadian infectious diseases and critical care physicians, multicentre retrospective study and BALANCE pilot RCT, all support the need for a randomized controlled trial comparing shorter (7 days) versus longer (14 days) antibiotic therapy for bloodstream infections. Prior to performing the main trial, Investigators completed a pilot trial in ICU patients to establish the feasibility of the research design, and to optimize the definitive trial. Investigators also completed a pilot trial of non-ICUs patients to test the feasibility, compare the patient population in two settings and to assess the reasonableness of expanding the main BALANCE Trial to non-ICU wards. The overall recruitment rate of the non-ICU ward pilot RCT exceeded the recruitment rate in the BALANCE ICU pilot RCT with a protocol adherence of 90%. The results of this pilot were used to estimate the necessary sample size recalculation, after merging the BALANCE ward trial with the BALANCE main trial, with the principle of maintaining an equal to smaller non-inferiority margin by the trial's completion. With the completion of this pilot RCT, the eligibility criteria for the BALANCE trial are also modified to broaden the inclusion of all bacteremic patients admitted to hospital. By defining the duration of treatment for bloodstream infections, BALANCE research program will help maximize the clinical cure of individual patients, while minimizing their risk of drug side effects, C. difficile, and antibiotic resistance. Since this intervention would require no new technology, and would reduce (rather than increase) health care costs, it would offer immediate benefits to patients and the healthcare system.

The BALANCE RCT will randomize hospitalized patients with bloodstream infection to 7 versus 14 days of adequate antibiotic treatment; the antibiotic drugs, doses, routes and interval will be left to the discretion of the treating team. Although placebo controls are not feasible, prolonged allocation concealment to day 7 will be used to mitigate selection bias. The primary analysis will assess whether 7 days is associated with non-inferior 90 day survival as compared to 14 days of treatment. Participants from the vanguard BALANCE pilot RCTs will be included in the BALANCE main RCT, and participating Canadian sites will continue to enrol patients. BALANCE international collaborators include New Zealand, Australia, Saudi Arabia, the United States, Israel and Switzerland.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is in ICU or non-ICU ward at the time the blood culture is drawn or reported as positive.
2. Patient has a positive blood culture with pathogenic bacteria.

Exclusion Criteria:

1. Patient already enrolled in the trial
2. Patient has severe immune system compromise, as defined by: absolute neutrophil count <0.5x109/L; or is receiving immunosuppressive treatment for solid organ or bone marrow or stem cell transplant
3. Patient has a prosthetic heart valve or synthetic endovascular graft (post major vessel repair with synthetic material) (note: coronary artery stents are not an exclusion)
4. Patient has documented or suspected syndrome with well-defined requirement for prolonged treatment:

   i) infective endocarditis; ii) osteomyelitis/septic arthritis; iii) undrainable/undrained abscess; iv) unremovable/unremoved prosthetic-associated infection (e.g. infected pacemaker, prosthetic joint infection, ventriculoperitoneal shunt infection etc.) (note: central venous catheters, including tunneled central intravenous catheter, and urinary catheters are not excluded unless the treating clinical team does not have equipoise for enrollment and randomization to either group)
5. Patient has a single positive blood culture with a common contaminant organism according to Clinical Laboratory & Standards Institute (CLSI) Guidelines: coagulase negative staphylococci; or Bacillus spp.; or Corynebacterium spp.; or Propionobacterium spp.; or Aerococcus spp.; or Micrococcus spp.
6. Patient has a positive blood culture with Staphylococcus aureus or Staphylococcus lugdunensis
7. Patient has a positive blood culture with Candida spp. or other fungal species.
8. Blood culture grows rare bacterial pathogens requiring prolonged treatment (e.g. Mycobacteria spp., Nocardia spp., Actinomyces spp., Brucella spp., Burkholderia pseudomallei)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3622 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
90 day survival | 90 days from index blood culture
  Survival at 90-days recorded as alive or dead at day 90 following index positive blood culture

SECONDARY OUTCOMES:
Hospital mortality | Expected average of 4 weeks assessed upto one year
  Recorded as alive or dead at hospital discharge following index positive blood culture
ICU mortality | Expected average of 2 weeks assessed upto one year
  Recorded as alive or dead at ICU discharge following index positive blood culture
Relapse rates of bacteremia with the same organism | Upto 30 days after adequate antibiotic treatment
  Defined as the recurrence of bacteremia due to original infecting organism (same Genus and species) after documentation of negative blood cultures or clinical improvement and within 30 days after completing course of adequate antimicrobial therapy.
Antibiotic allergy and adverse events | Upto 30 days from start of antibiotic treatment
  Effect of medication on body that produces the allergic reaction to a medication like:
  * Hives
  * Itching of the skin or eyes
  * Skin rash
  * Swelling of the lips, tongue, or face
  * Wheezing
  * Organ toxicity
Rates of C. difficile infection in hospital | Upto 30 days after index blood culture collection date
  Defined as a positive PCR or ELISA test for Clostridium difficile toxin in the context of diarrhea within hospital of bacteremia diagnosis.
Rates of secondary nosocomial infection/colonization with antimicrobial resistant organisms in hospital | Upto 30 days after index blood culture collection date
  Colonized or infected with at least one highly-resistant microorganism during their hospital stay
ICU length of stay | Expected for an average of 30 days assessed up to 1 year
  Defined as the duration between index blood culture and discharge from the ICU for a consecutive 48-hour period
Hospital length of stay | Expected for an average of 30 days assessed up to 1 year
  Defined as the duration between index blood culture and discharge date from hospital
Mechanical ventilation duration | Expected for an average of 30 days
  Defined as the number of consecutive days receiving invasive (via an endotracheal tube or tracheostomy), or non-invasive (via a facemask, nasal mask, or helmet) ventilation
Antibiotic free days | Upto 30 days after adequate antibiotic treatment
  Defined as the number of days during the 28 days after the start of adequate antibiotics in which patients did not receive any antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (68):
- United States (2):
  - NYU School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Australia (17):
  - Bankstown Hospital, Bankstown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital ICU, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Ballarat Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Casey Hospital, Berwick, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital- Monash Health, Dandenong, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Peninsula Private Hospital, Langwarrin, Victoria
  - Cabrini Health, Malvern, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Hospital, Subiaco, Western Australia
- Canada (37):
  - Foothills Hospital, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Lions Gate Hospital, Vancouver, British Columbia
  - Royal Columbian Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Island Health, Victoria, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - William Osler Health System, Brampton, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Brantford General Hospital, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Hospitalier Régional de Trois-Rivières, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - Royal Victoria Hospital, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Israel (2):
  - Rabin Medical Center, Petah Tikva, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky, Tel Aviv
- New Zealand (7):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Taranaki Hospital, New Plymouth
  - Rotorua Hospital, Rotorua
  - Wellington Hospital, Wellington
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre, Jeddah
  - King Abdulaziz Medical City, Riyadh
- University hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong SWX, Pinto R, Rishu A, Tong SYC, Commons RJ, Conly JM, Evans GA, Fralick M, Kandel C, Lagace-Wiens PRS, Lee TC, Lother SA, MacFadden DR, Marshall JC, Martel-Laferriere V, Mayette M, McDonald EG, Neary JD, Prazak J, Raby E, Regli A, Rogers BA, Smith S, Taggart LR, Wang HT, Wuerz T, Yahav D, Young PJ, Fowler RA, Daneman N; BALANCE trial consortium. Identifying heterogeneity of treatment effect for antibiotic duration in bloodstream infection: an exploratory post-hoc analysis of the BALANCE randomised clinical trial. EClinicalMedicine. 2025 Apr 10;83:103195. doi: 10.1016/j.eclinm.2025.103195. eCollection 2025 May. PMID 40256773
- [Derived] BALANCE Investigators, for the Canadian Critical Care Trials Group, the Association of Medical Microbiology and Infectious Disease Canada Clinical Research Network, the Australian and New Zealand Intensive Care Society Clinical Trials Group, and the Australasian Society for Infectious Diseases Clinical Research Network; Daneman N, Rishu A, Pinto R, Rogers BA, Shehabi Y, Parke R, Cook D, Arabi Y, Muscedere J, Reynolds S, Hall R, Dwivedi DB, McArthur C, McGuinness S, Yahav D, Coburn B, Geagea A, Das P, Shin P, Detsky M, Morris A, Fralick M, Powis JE, Kandel C, Sligl W, Bagshaw SM, Singhal N, Belley-Cote E, Whitlock R, Khwaja K, Morpeth S, Kazemi A, Williams A, MacFadden DR, McIntyre L, Tsang J, Lamontagne F, Carignan A, Marshall J, Friedrich JO, Cirone R, Downing M, Graham C, Davis J, Duan E, Neary J, Evans G, Alraddadi B, Al Johani S, Martin C, Elsayed S, Ball I, Lauzier F, Turgeon A, Stelfox HT, Conly J, McDonald EG, Lee TC, Sullivan R, Grant J, Kagan I, Young P, Lawrence C, O'Callaghan K, Eustace M, Choong K, Aslanian P, Buehner U, Havey T, Binnie A, Prazak J, Reeve B, Litton E, Lother S, Kumar A, Zarychanski R, Hoffman T, Paterson D, Daley P, Commons RJ, Charbonney E, Naud JF, Roberts S, Tiruvoipati R, Gupta S, Wood G, Shum O, Miyakis S, Dodek P, Kwok C, Fowler RA; The BALANCE Investigators, for the Canadian Critical Care Trials Group, the Association of Medical Microbiology and Infectious Disease Canada Clinical Research Network, the Australian and New Zealand Intensive Care Society Clinical Trials Group, and the Australasian Society for Infectious Diseases Clinical Research Network. Antibiotic Treatment for 7 versus 14 Days in Patients with Bloodstream Infections. N Engl J Med. 2025 Mar 13;392(11):1065-1078. doi: 10.1056/NEJMoa2404991. Epub 2024 Nov 20. PMID 39565030
- [Derived] Rogers BA, Fowler R, Harris PNA, Davis JS, Pinto RL, Bhatia Dwivedi D, Rishu A, Shehabi Y, Daneman N. Non-inferiority trial of a shorter (7 days) compared with a longer (14 days) duration of antimicrobial therapy for the treatment of bacteraemic urinary sepsis, measured by microbiological success after the completion of therapy: a substudy protocol for the Bacteraemia Antibiotic Length Actually Needed for Clinical Effectiveness (BALANCE) multicentre randomised controlled trial. BMJ Open. 2023 Jun 26;13(6):e069708. doi: 10.1136/bmjopen-2022-069708. PMID 37369422
- [Derived] Daneman N, Rishu AH, Pinto RL, Arabi YM, Cook DJ, Hall R, McGuinness S, Muscedere J, Parke R, Reynolds S, Rogers B, Shehabi Y, Fowler RA; Canadian Critical Care Trials Group. Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness (BALANCE) randomised clinical trial: study protocol. BMJ Open. 2020 May 11;10(5):e038300. doi: 10.1136/bmjopen-2020-038300. PMID 32398341